CLINICAL TRIAL: NCT05940493
Title: A Phase 2 Multicenter, Double-blind, Randomized-controlled Study of Abemaciclib (CDK4 and 6 Inhibitor) in Newly Diagnosed RB-proficient Grade 3 Meningioma Participants
Brief Title: Abemaciclib in Newly Diagnosed Meningioma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nader Sanai (Other)
Collaborators: Eli Lilly and Company (Industry); Barrow Neurological Institute (Other); Ivy Brain Tumor Center (Other)
Responsible Party: Sponsor-Investigator, Nader Sanai, Chief Scientific Officer/Director of the Ivy Brain Tumor Center, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-14; 23-500-352-34-38 (Other: St. Joseph's Hospital)
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-02

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — abemaciclib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All site study personnel, except the unblinded dispenser and verifier, will be aware of whether participants are receiving abemaciclib or placebo until the study is formally unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment (Abemaciclib) (Experimental): Administered twice daily on days 1-28 of each 28-day cycle.
  Interventions: Drug: Abemaciclib
- Placebo (Placebo Comparator): Administered twice daily on days 1-28 of each 28-day cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abemaciclib — Tablet
  Arms: Active Treatment (Abemaciclib)
Drug: Placebo — Tablet
  Other Names: Abemaciclib placebo
  Arms: Placebo

SUMMARY:
This study is being done to learn about how an investigational drug called abemaciclib works in treating patients with a newly-diagnosed grade 3 meningioma. Abemaciclib is a drug that is approved by the FDA, but not for brain tumors.

Participants who consent to the trial will have surgical tissue collected from the planned surgical resection and tested. If the tissue shows positive results for RB cells and participants are qualified, they will be enrolled and receive study treatment two to five weeks after completing standard-of-care radiation therapy.

This is a randomized clinical trial which means that participants will be randomly assigned to a treatment based on chance, like a flip of a coin. Neither the participant nor the researcher chooses the assigned group. Randomization will help the researchers study how the drug works by comparing the difference between the study drug and the placebo and how they work in treating brain tumors. This is a double-blinded study, which means that neither the participant nor the study team will know which treatment the participant is receiving.

ELIGIBILITY:
Inclusion Criteria:

* Participants with newly diagnosed intracranial WHO Grade 3 meningioma; or,
* Participants with previous lower grade meningioma and histopathologically confirmed newly transformation to Grade 3.
* Plan to receive or have received upfront standard of care radiation therapy (RT) for the newly diagnosed WHO Grade 3 meningioma.
* No prior treatment for Grade 3 meningioma other than surgical resection or biopsy and upfront RT. If previously diagnosed with a lower grade meningioma, no prior treatment other than surgical resection or biopsy and no prior RT.
* Ability to understand and the willingness to sign a written informed consent document (personally or by the legally authorized representative, if applicable).
* Participant has voluntarily agreed to participate by giving written informed consent (personally or via legally authorized representative[s], and assent, if applicable). Written informed consent for the protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally document and witnessed, ideally via an independent trusted witness. Participant must be willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures.
* Age ≥18 years at time of consent.
* Have a performance status (PS) of ≤2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Ability to swallow oral medications.
* Participant has adequate bone marrow and organ function as defined by the following laboratory values (as assessed by the local laboratory for eligibility):

  * Adequate Bone Marrow Function: absolute neutrophil count ≥1,500/mcL, platelets ≥100,000/mcL, and hemoglobin ≥8.0 g/dL (individual may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator; initial treatment must no begin earlier than the day after any erythrocyte transfusion).
  * Adequate Hepatic Function: total bilirubin ≤1.5x ULN (individuals with Gilbert's syndrome with a total bilirubin ≤2.0x ULN and direct bilirubin within normal limits are permitted), AST/SGOT ≤3x ULN, and ALT/SGPT ≤3x ULN.
* Confirmed negative serum pregnancy test (β-hCG) before starting study treatment or participant who is no longer of childbearing potential due to surgical, chemical, or natural menopause.
* For females of reproductive potential: use of highly effective contraception during study participation and for an additional 3 weeks after the end of treatment administration.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner and for an additional 3 weeks after the end of treatment administration.

Exclusion Criteria:

* Prior history of cancer with ongoing treatment of disease.
* Pregnancy or breastfeeding.
* Known allergic reactions to components of the abemaciclib.
* Active infection or fever >38.5°C requiring systemic antibiotic, antifungal or antiviral therapy within 4 weeks of Day 1.
* Known to have active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis.
* Known active systemic bacterial infection (requiring IV antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known HIV positivity or with known HBV or HCV). Screening is not required for enrollment.
* Participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
* Prior therapy with any CDK4/6 inhibitor. Prior therapy is defined as therapeutic dosing.
* Treatment with another investigational drug within 5 half-lives of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 months
  Progression free survival (PFS24) rate measured from the time of surgery to date of recurrence

SECONDARY OUTCOMES:
Drug-related toxicity | Up to 30 days after last study dose
  Incidence of drug-related toxicity
Adverse Events | Up to 30 days after last study dose
  Number of adverse events through study completion
Deaths | 24 months
  Number and incidence of deaths
Incidence of clinical laboratory abnormalities per CTCAE | Up to 30 days after last study dose
  Clinical laboratory abnormalities per CTCAE
Progression-free survival in participants | 12 months
  12 month progression-free survival (PFS12) rate measured from the time of surgery to date of recurrence.
Overall Survival | 24 months
  Overall survival at 24 months
Median Overall Survival | 5 years
  Median overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Principal Investigator — Ivy Brain Tumor Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No